CLINICAL TRIAL: NCT04114851
Title: The Effects of Objective Estimation of Pain Response With Person-centered Care in Patients Undergoing Endoscopic Surgery (FESS, Concaplasty or Lateral Rhinotomy)
Brief Title: The Effects of Objective Estimation of Pain Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-01023
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia; Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Investigator
Masking Description: control group will be masked so that the monitor index will not be seen by the caregiver/investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Patients who get active monitor NoL
  Interventions: Device: NoL
- control (No Intervention): control no NoL

INTERVENTIONS:
Device: NoL — NoL active
  Arms: Active

SUMMARY:
There are different types of pain generators that give different pain symptoms. In anesthesia and surgery, the pain generator in connection with, for example, surgical procedures is referred to as nociceptive pain. However, there is not enough evidence to support that these physiological changes are direct signs of nociceptive stimulation. The same changes can be seen with an autonomous stress trigger of origin other than just nociceptive stimulation. This means that healthcare professionals who provide anesthesia to patients during, for example, surgery may provide unnecessary pain relief drugs or do not provide pain relief when needed. This is also true in awake patients when pain is complex that, for example, concerns may increase the experience of pain and that healthcare professionals may even then misinterpret and provide more pain-relieving drugs despite the actual need for another drug or complementary treatment.

Examples of these include heart rate variation, specific patterns in blood pressure and heart rate response, heart rate amplitude, heart rate range, skin sweating and pupil response. The reason why these changes have not been used to interpret nociceptive stimulation is directly linked to an absence of technology that makes it possible to collect data and interpret these changes.

list a number of methods / techniques that are under development, one of which is the Nociception Level Index (NoL). NoL is an indexed value between 0 and 100 and is based on a non-linear combination of nociception-related physiological variables (including heart rate variation, plethysmograph pulse wave amplitude (PPGA) and changes in skin resistance). Possibly NoL is the first evidence-based clinical technology that can discriminate pain response when physiological response is not measured.

The research field in the area of non-invasive objective monitoring of pain response in relation to patients' experience of pain is currently almost non-existent in anesthesia / anesthesia care This in turn can also lead to the development of patient safety both during anesthesia and after surgery at nursing department for example, patient-controlled and epidural pain relief in postoperative pain care. investigators intend to study the variation of the NoL index linked to the need for opioids during anesthesia and also after completed anesthesia when the patient wakes up and is in the ward.

DETAILED DESCRIPTION:
Investigators study patients undergoing functional endoscopic sinus surgery (FESS), concaplasty or lateral rhinotomy and who receive routine general anesthesia (anesthesia). These patients often have an age between 30-60 years and not infrequently assessed with regard to intraoperative and postoperative pain response. During the anesthesia study and after anesthesia, an equipment that monitors the pain response NoL (pain monitor) is used.

This kind of pain monitor has been around for about 10 years. Over the past 5 years, its technology has evolved so much that in various countries it has become a monitoring system that is used as a complement to anesthesia.

The study will be a randomized intervention study in which the random determines whether the patient's pain level is monitored using NoL or only according to traditional clinical assessment intra- and post-operatively. The patient will be assessed with the post-Qrs test, partly preoperatively (baseline) and partly post-operatively to assess the rate of recovery compared to baseline. The collected data is analyzed afterwards to possibly determine whether it is possible to determine differences in recovery, based on choice of pain monitoring method (Pain NoL or clinical assessment, pulse, blood pressure, BIS index, NoL index, amount of opioid intraoperatively and opioid amount postoperatively, VAS / NRS).

Patients included in the study will be persons over the age of 18 and who agree to participate. Both women and men are included. Exclusion criteria include problems with the Swedish language or other communicative difficulties that make the assessment more difficult and patients with pacemakers.

Both groups are anesthetized with propofol infusion and oxygen in the air, which is given analgesic remifentanil during surgery.

Randomization is done through mixed, closed envelopes. Prior to the anesthesia, extra oxygen will be added and standard monitoring will be connected to the patient (ECG, noninvasive blood pressure measurement, saturation, NMT, NoL).

Form, Postop-QRS test, with questions will be reviewed with the patient the day before or the same day as the surgery and postoperatively. The tests are intended to measure alertness, pain, nausea, vomiting and cognitive function and general recovery.

The BIS index, NoL index, heart rate, blood pressure and saturation are regularly measured and recorded in special protocol. (NoL blinded, these index values are stored directly from the monitor on a so-called USB memory stick)

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 yrs old

Exclusion Criteria: Cognitive decline, mental illness, drug addicts and non-Swedish speakers. Skin damage to fingers that make application more difficult.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Amount of opioid used | 24 hours
  Amount of opioid used

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University hospital, Gothenburg, Sweden